CLINICAL TRIAL: NCT03786406
Title: A Non-interventional Cross-sectional Study to Capture the Prevalence of Cardiovascular Disease in Patients With Type 2 Diabetes in Selected Countries in Europe
Brief Title: An International Survey of the Occurrence of Diseases That Affects the Heart and Blood Vessels Among People With Type 2 Diabetes
Acronym: EU-CAPTURE
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN2211-4423; U1111-1207-2816 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-12-20; First posted 2018-12-26 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- T2DM patients seen in routine practice: All anti-diabetic and cardiovascular (CV) medication will be prescribed at the physician's discretion under routine clinical practice conditions.
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No specific intervention is studied. All anti-diabetic and CV medication will be prescribed at the physician's discretion under routine clinical practice conditions.

SUMMARY:
The purpose of the study is to register the occurrence of cardiovascular disease among type 2 diabetes (T2DM) patients across five selected countries in Europe. Participants will be asked to give information about their health. Participants will continue their normal way of life and will not get any medication other than what has been prescribed to them by their doctor. Participants' participation will be one day/one visit at study doctor. The study will last for about 3 months in total.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained before any study-related activities (study-related activities are any procedures related to recording of data according to protocol)
* Male or female, age greater than or equal to 18 years at the time of signing informed consent
* Diagnosed with type 2 diabetes mellitus greater than or equal to 180 days prior to the day of signing the informed consent

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study
* Diagnosed with Type 1 diabetes
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Patients with known congenital heart disease/malformation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of male and female adults diagnosed with (type 2 diabetes mellitus (T2DM).
Sampling Method: Non-Probability Sample
Enrollment: 2275 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Diagnosed with cerebrovascular disease: Ischaemic stroke, haemorrhagic stroke, stroke (unspecified) and/or transient ischaemic attack | Day 1
  Percentage of participants (Y/N).
Diagnosed with CVD: Myocardial infarction, stable coronary artery disease (SCAD) also referred as angina (pectoris), other ischaemic heart disease and/or past revascularisation procedures | Day 1
  Percentage of participants (Y/N).
Diagnosed with symptomatic heart failure: New York Heart Association Functional Classification (NYHA) (group IIIV) and/or left ventricular ejection fraction (LVEF) greater than or equal to 50 percent, LVEF 40-49 percent and LVEF less than 40 percent) | Day 1
  Percentage of participants (Y/N).
Diagnosed with asymptomatic heart failure | Day 1
  Percentage of participants (Y/N).
Hospitalisation for heart failure | Day 1
  Percentage of participants (Y/N).
Diagnosed with cardiac arrhythmia: Atrial fibrillation or flutter, ventricular tachycardia and/or ventricular fibrillation | Day 1
  Percentage of participants (Y/N).
Diagnosed with aortic diseases: Aortic dissection, aortic aneurysms and/or thromboembolic aortic disease | Day 1
  Percentage of participants (Y/N).
Diagnosed with peripheral artery disease: Asymptomatic peripheral arterial disease (PAD) defined as Low Ankle-Brachial Index (less than 0.90) or pulse abolition, claudication, limb ischemia and/or non-traumatic amputation | Day 1
  Percentage of participants (Y/N).
Diagnosed with carotid artery disease | Day 1
  Percentage of participants (Y/N).

SECONDARY OUTCOMES:
High risk of CVD (above 20% over 10 years) according to the risk engine from the United Kingdom Prospective Diabetes Study (UKPDS) | Day 1
  Percentage of participants (Y/N).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (40):
- Czechia (12):
  - Novo Nordisk Investigational Site, Benátky nad Jizerou
  - Novo Nordisk Investigational Site, Boskovice
  - Novo Nordisk Investigational Site, Brandýs nad Labem
  - Novo Nordisk Investigational Site, Břeclav
  - Novo Nordisk Investigational Site, Chomutov
  - Novo Nordisk Investigational Site, Hradec Králové
  - Novo Nordisk Investigational Site, Kroměříž
  - Novo Nordisk Investigational Site, Olomouc
  - Novo Nordisk Investigational Site, Orlová
  - Novo Nordisk Investigational Site, Ostrava
  - Novo Nordisk Investigational Site, Pilsen
  - Novo Nordisk Investigational Site, Prague
- France (10):
  - Novo Nordisk Investigational Site, Chartres
  - Novo Nordisk Investigational Site, Courpière
  - Novo Nordisk Investigational Site, Le Creusot
  - Novo Nordisk Investigational Site, Lyon
  - Novo Nordisk Investigational Site, Montélimar
  - Novo Nordisk Investigational Site, Saint-Saëns
  - Novo Nordisk Investigational Site, Sathonay-Camp
  - Novo Nordisk Investigational Site, Strasbourg
  - Novo Nordisk Investigational Site, Tarare
  - Novo Nordisk Investigational Site, Vénissieux
- Italy (18):
  - Novo Nordisk Investigational Site, Albano Laziale
  - Novo Nordisk Investigational Site, Ariano Irpino
  - Novo Nordisk Investigational Site, Bagno a Ripoli
  - Novo Nordisk Investigational Site, Brindisi
  - Novo Nordisk Investigational Site, Catanzaro
  - Novo Nordisk Investigational Site, Fano
  - Novo Nordisk Investigational Site, Ferrara
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Messina
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Napoli
  - Novo Nordisk Investigational Site, Negrar (VR)
  - Novo Nordisk Investigational Site, Orvieto
  - Novo Nordisk Investigational Site, Partinico (PA)
  - Novo Nordisk Investigational Site, Ravenna
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, Rozzano (MI)
  - Novo Nordisk Investigational Site, Savigliano (CN)

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://www.novonordisk-trials.com

REFERENCES:
- [Result] Mosenzon O, Alguwaihes A, Leon JLA, Bayram F, Darmon P, Davis TME, Dieuzeide G, Eriksen KT, Hong T, Kaltoft MS, Lengyel C, Rhee NA, Russo GT, Shirabe S, Urbancova K, Vencio S; CAPTURE Study Investigators. CAPTURE: a multinational, cross-sectional study of cardiovascular disease prevalence in adults with type 2 diabetes across 13 countries. Cardiovasc Diabetol. 2021 Jul 27;20(1):154. doi: 10.1186/s12933-021-01344-0. PMID 34315481
- [Derived] Vencio S, Vianna AGD, da Silva MACF, Precoma DB. Contemporary (2019) prevalence of cardiovascular disease in adults with type 2 diabetes in Brazil: the cross-sectional CAPTURE study. Diabetol Metab Syndr. 2022 Jan 10;14(1):5. doi: 10.1186/s13098-021-00775-9. PMID 35012646